CLINICAL TRIAL: NCT02410863
Title: Biopsy- and Biology-driven Optimization of Targeted Therapy of Metastatic Melanoma in BRAF Inhibitor Non-pretreated and Pretreated Subjects With Advanced, Non-resectable (STAGE IIIC) or Metastatic (StAGE IV) BRAF Mutation-positive Melanoma
Brief Title: Biopsy- and Biology-driven Optimization of Targeted Therapy in Subjects With Advanced Melanoma
Acronym: BOTTOM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of recruitment due to changed therapy options
Sponsor: Prof. Dr. med. Dirk Schadendorf (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Dirk Schadendorf, Sponsor-Investigator, University Hospital, Essen
Organization: University Hospital, Essen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bottom_2012
Record Dates: First submitted 2015-04-02; First posted 2015-04-08 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Malignant Melanoma
Keywords: Stage III or IV with BRAF V600E/K mutation
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (BRAFi naïve) (Experimental): Dabrafenib (BRAFi) and trametinib (MEKi) will be administered orally at their recommended doses for combination therapy of 150 mg twice daily (BID) and 2 mg daily.
  Interventions: Drug: Dabrafenib; Drug: Trametinib
- Cohort B (BRAFi / MEKi rechallenge) (Experimental): Dabrafenib (BRAFi) and trametinib (MEKi) will be administered orally at their recommended doses for combination therapy of 150 mg twice daily (BID) and 2 mg daily
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — 150 mg twice daily
  Other Names: Tafinlar
Drug: Trametinib — 2 mg daily
  Other Names: Mekinist

SUMMARY:
This is an open-label, multi-center, clinical phase II study to explore the correlation of the genetic make-up of the treated tumor before start of therapy and to correlate clinical response at 8 weeks as well as metabolic response at 2 and 8 weeks with genetic features of the tumor.

It will be conducted as a rationale optimization of targeted therapy in BRAF naïve and pretreated patients.

Prerequisite for all patients is the availability of tumor sample at start of treatment in order to determine the underlying driver mutation (BRAF mutational status) as well as molecular composition by next generation sequencing (NGS) and assessable lesions for biopsy at week 2. Melanoma patients in stage III (non-resectable) and stage IV are sorted into Cohort A or B according to their previous BRAF-treatment and treated with dabrafenib and trametinib (cohort A and B)

DETAILED DESCRIPTION:
In this open-label, multi-center, clinical phase II study melanoma patients in stage III (non-resectable) and stage IV are sorted into Cohort A or B according to their previous BRAF-treatment:

Cohort A (BRAFi naïve): Patients who have not received prior BRAFi or MEKi-therapy. Dabrafenib (BRAFi) and trametinib (MEKi) will be administered orally at their recommended doses for combination therapy of 150 mg twice daily (BID) and 2 mg daily (QD). Clinical endpoint is clinical response at week 8. Metabolic response will be assessed at week 2 and 8. Treatment will continue until disease progression, death, unacceptable toxicity, or withdrawal of consent.

Cohort B (BRAFi / MEKi rechallenge): Patients with CR/PR as best response to previous BRAFi / MEKi combination therapy, discontinuation of this therapy after progression and different therapy for > 3 months prior to enrollment.

These patients will receive dabrafenib and trametinib at their recommended combination therapy doses of 150 mg twice daily (BID) and 2 mg daily (QD).

Treatment will continue until disease progression, death, unacceptable toxicity, or withdrawal of consent.

Survival will be assessed every 3 months after the final dose of BRAFi / MEKi until the end of the follow-up phase for the individual patient.

Follow up phase for each subject is 1 year following first treatment dose. End of study will be at recruitment finished plus 1 year post start of treatment of last patient thus ensuring that 1 year survival rate can be estimated.

Biopsies taken before start of treatment, after 2 weeks (+/- 4 days) and after progressive disease will be analyzed by Next generation sequencing (NGS), immunohistochemistry (IHC), phosphorplex Luminex as well as by reverse phase protein array in order to determine the magnitude of suppression of downstream signaling as well as reactivation of adaptative mechanisms.

Rebiopsy is mandatory after 2 weeks and in case of progressive disease in order to determine mechanisms of adaptation of the signaling pathway downstream.

The experimental molecular data will be analyzed in correlation with clinical response at week 8 (defined as partial or complete response according to RECIST) and metabolic responses at weeks 2 and 8 (responders are defined as those patients with changes of >66% in the Standard Uptake value (SUVmax) between interim PET and baseline PET.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. Signed written informed consent.
3. Histologically confirmed cutaneous melanoma that is either Stage IIIc (unresectable) or Stage IV (metastatic), and determined to be BRAF V600E/K mutation-positive by the central laboratory. Subjects with ocular or mucosal melanoma are not eligible.
4. Assessable lesion for biopsy at week 2 not inferring with RECIST measurements (Biopsies for genetic/biomarker analyses must be taken from lesions not required for disease assessment)
5. Measurable disease, i.e., present with at least one measurable lesion per RECIST, version 1.1 for the definition of a measureable lesion.
6. For Cohort A: Must NOT have received prior treatment with BRAF or MEK inhibitor.

   If a prior systemic therapy (such as but not limited to chemotherapy, immunotherapy, biologic, vaccine and/or investigational treatment) in metastatic disease has been administered, four weeks or more since last systemic treatment must have passed. Must have recovered from any acute toxicity associated with prior therapy.
7. For Cohort B: Must have shown PR/CR during treatment with selective BRAF/MEK combination treatment that was discontinued due to tumor progression and received subsequent alternative treatment (such as but not limited to surgery, chemotherapy, immunotherapy, biologic, vaccine and/or investigational treatment), with a period of at least 3 months since last intake of BRAF/MEK inhibitor
8. All prior treatment-related toxicities (except alopecia) must be ≤ Grade 1 according to the Common Terminology Criteria of Adverse Events (CTCAE, Version 9. Able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.

10. Women of childbearing potential must have a negative urin pregnancy test within 7 days prior to registration and agree to use effective contraception, as defined in Section 9.8 throughout the treatment period, and for 4 months after the last dose of study treatment.

Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception as described in Section 9.8 throughout the treatment period, and for 4 months after the last dose of study treatment. 11. An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 12. Adequate baseline organ function defined as Absolute Neutrophil Count ≥1.2 × 109/L Hemoglobin ≥ 9 g/dL Platelet count ≥ 100 x 109/L Prothrombinzeit (PT/INR) and Partial thromboplastin time ≤ 1.3 x upper laboratory norm (ULN) Albumin ≥ 2.5 g/dL Total bilirubin ≤ 1.5 x ULN Aspartate aminotransferase and Alanine Aminotransferase ≤ 2.5 x ULN Serum creatinine ≤ 1.5 mg/dL 13. A left ventricular ejection fraction (LVEF) ≥ the institutional lower limit of normal as measured by ECHO

Exclusion Criteria:

1. Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 21 days prior to registration and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to registration.
2. Taken an investigational drug within 28 days or 5 half-lives (minimum 14 days), whichever is shorter, prior to registration.
3. Current use of a prohibited medication
4. History of another malignancy. Exception: Subjects who have been disease-free for 3 years, subjects with a history of completely resected non-melanoma skin cancer, and/or subjects with successfully treated in situ carcinoma are eligible. Subjects with second malignancies that are indolent or definitively treated may be enrolled.
5. Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the subject's safety, obtaining informed consent, or compliance with study procedures.
6. Known Human Immunodeficiency Virus (HIV), active Hepatitis B Virus (HBV), or active Hepatitis C Virus (HCV). Subjects with chronic or cleared HBV and/or HCV are eligible.
7. A history of glucose-6-phosphate dehydrogenase (G6PD) deficiency.
8. Subjects with brain metastases are excluded, unless:

   * All known lesions must be previously treated with surgery or stereotactic radiosurgery, and
   * Brain lesion(s), if present, must be confirmed stable (ie, no increase in lesion size) for 90 days prior to first dose of study drug(s). This must be documented with two consecutive MRI or CT scans using contrast, and
   * Asymptomatic with no corticosteroids requirement for 30 days prior to first dose of study drug(s), and
   * No enzyme-inducing anticonvulsants for 30 days prior to first dose of study drug(s).

   In addition, even in cases of no evidence of disease (NED), confirmation on two consecutive MRI or CT scans using contrast will be required. Enrollment of a subject with brain metastases who meet the above criteria requires approval of the sponsor
9. A history or evidence of cardiovascular risk including any of the following:

   1. A QT interval corrected for heart rate using the Bazett's formula (QTcB; ³ 480 msec;
   2. A history or evidence of current clinically significant uncontrolled arrhythmias; Exception: Subjects with controlled atrial fibrillation for > 30 days prior to registration are eligible.
   3. A history of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within 6 months prior to registration; or
   4. A history or evidence of current ≥ Class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines.
10. A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR) including:

    Presence of predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled hypertension, uncontrolled diabetes mellitus, or a history of hyperviscosity or hypercoagulability syndromes); or

    Visible retinal pathology as assessed by ophthalmic examination that is considered a risk factor for RVO or CSR such as:

    i. Evidence of new optic disc cupping; ii. Evidence of new visual field defects on automated perimetry; iii. Intraocular pressure > 21 mmHg as measured by tonography.
11. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO).
12. Interstitial lung disease or pneumonitis
13. Pregnant or breast-feeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Correlation of clinical response at week 8 of targeted therapy with molecular results of the biopsies. | Week 8
  To broaden the understanding of molecular characterization of the melanoma in correlation to the clinical response (defined as partial or complete response according to RECIST) at week 8 of targeted therapy in different pre-treated patients with advanced/metastatic BRAF V600E/K mutation-positive cutaneous melanoma.

SECONDARY OUTCOMES:
Correlation of the tumor´s molecular composition to metabolic responses | Baseline, week 2 and 8
  To correlate the tumor´s molecular composition to metabolic responses and biological effects on the downstream signaling cascade in order to get first insights into an adaptive mechanism in the downstream signaling of an oncogenic driver mutation upon its selective inhibition.
Safety / toxicity according to the Common Toxicity Criteria (CTC, Version 4.0) | 1 year
  Occurrence of adverse events and reactions
Progression free survival rate | 6 and 12 months
  Proportion of patients with PFS after date of the first dose of study medication until the first documented tumor progression date or date of death, whichever occurs first.
Overall survival | 6 and 12 months
  Time after date of the first dose of study medication until documented date of death
Progression free survival according to RECIST criteria | 6 and 12 months
  Time after date of the first dose of study medication until the first documented tumor progression date or date of death, whichever occurs
Overall response rate according to RECIST criteria | 6 and 12 months
  Proportion of patients with PR and CR
Disease control rate according to RECIST criteria | 6 and 12 months
  Proportion of patients with SD, PR and CR

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Schadendorf, Prof. Dr., Principal Investigator — University Hospital, Essen
Locations (6):
- Germany (6):
  - National Centre for Tumour Diseases (NCT), Heidelberg, Baden-Wurttemberg
  - University Hospital Tübingen, Tübingen, Baden-Wurttemberg
  - Elbe Kliniken Stade - Buxtehude GmbH, Clinic for Dermatology, Buxtehude, Lower Saxony
  - University Hospital Essen, Essen, North Rhine-Westphalia
  - University Hospital Mainz, Clinic for Dermatology, Mainz, Rhineland-Palatinate
  - Universitätsklinik Carl Gustav Carus der Technischen Universität Dresden, Dresden, Saxony